CLINICAL TRIAL: NCT01176773
Title: Safety and Effectiveness of Juvéderm® Ultra Lip Injectable Gel for Lip Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: S15-002
Record Dates: First submitted 2010-03-23; First posted 2010-08-06 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2013-12

CONDITIONS: Lip Enhancement

ARMS (1):
- Juvéderm® Ultra Lip Injectable Gel (Experimental)
  Interventions: Device: hyaluronic acid gel

INTERVENTIONS:
Device: hyaluronic acid gel — Dosage per Investigator's discretion to obtain lip treatment goal; 1 touch-up treatment is allowed 14 days after initial treatment. Maximum total volume per subject is 2.0 mL

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of Juvéderm® Ultra Lip Injectable Gel for lip enhancement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Desire enhancement of his/her vermilion borders and/or vermilion mucosa Cupid's bow, philtral columns, perioral lines, and oral commissures may also be treated
* Have a baseline score of Minimal of Mild, as assessed by the Investigator according to the 4-point Lip Fullness Scale (Minimal, Mild, Moderate, Marked)
* Have established a realistic Lip Fullness treatment goal that Investigator agrees is achievable

Exclusion Criteria:

* Have undergone cosmetic facial, lip or perioral procedures [e.g., face-lift or other surgeries which may alter the appearance of the lips or perioral area (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures), tissue augmentation with dermal fillers or fat injections, or mesotherapy] anywhere in the face or neck, or BOTOX® Cosmetic injections in the lower face (below the orbital rim), within 6 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study. Note: Prior treatment with Hyaluronic Acid fillers and/or collage is allowed, provided the treatment was administered not less than 6 months prior to study entry
* Have ever received semi-permanent fillers or permanent facial implants (e.g., calcium hydroxylapatite, L-polylactic acid, PMMA, silicone, ePTFE) anywhere in the lips, or be planning to be implanted with any of these products at any time during the study
* Have a history of anaphylaxis, multiple severe allergies, atopy, allergy to local anaesthesia agents, hyaluronic acid products or Streptococcal protein, or be planning to undergo desensitization therapy during the term of the study
* Are pregnant, lactating, or planning to become pregnant at any time during the study
* Have received investigational product within 30 days prior to study enrollment or be planning to participate in another investigation during the course of this study
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
* Have a history of or currently suffer from autoimmune disease
* Have a history of treatment with interferon for chronic hepatitis C
* Be on an ongoing regimen of anti-coagulation therapy (e.g., warfarin) or have taken NSAIDs (e.g. aspirin, ibuprofen) or other substances known to increase coagulation time (e.g. herbal supplements with garlic or Gingko Biloba) within 10 days of undergoing study device injection. Note: Study device injection may be delayed as necessary to accommodate this 10-day wash out period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Belfast
  - Cheadle
  - Halesowen
  - Sutton Coldfield

REFERENCES:
- [Background] Eccleston D, Murphy DK. Juvederm((R)) Volbella in the perioral area: a 12-month prospective, multicenter, open-label study. Clin Cosmet Investig Dermatol. 2012;5:167-72. doi: 10.2147/CCID.S35800. Epub 2012 Oct 26. PMID 23152693

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Started | 62
Completed | 59
Not Completed | 3
Not completed — Screen Failure | 2
Not completed — Withdrew consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 60

OUTCOME MEASURES:

1. Primary Outcome: Investigator Assessment of the Subject's Overall Lip Fullness on the 4-point Lip Fullness Scale
Description: The responder rate at 3 months, where a responder was defined as an improvement (increase) on the Lip Fullness Scale of ≥ 1 grade compared with the baseline assessment
Time Frame: 3 months
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- Juvéderm® Ultra Lip Injectable Gel: The Investigator determined the appropriate volume to inject based on clinical experience and the subject's cosmetic goals for lip enhancement.
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Number analyzed (Participants) | 59
percentage of responders | 93.2 [83.54 to 98.12]

2. Secondary Outcome: Investigator Assessment of Perioral Line Severity Using the Perioral Line Severity Scale
Description: Score on 4-point Perioral Line Severity Scale, where 0 is none and 3 is severe. A decreased score indicates improvement.
Time Frame: 12 months
Population: All subjects who were treated for perioral lines
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Number analyzed (Participants) | 26
units on a scale | 1.5 (0.69)

3. Secondary Outcome: Investigator Assessment of Oral Commissures Using the Oral Commissures Severity Scale
Description: Score on 4-point Oral Commissures Severity Scale, where 0 is none and 3 is severe. A decreased score indicates improvement.
Time Frame: 12 months
Population: All subjects who were treated in their oral commissures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Number analyzed (Participants) | 52
units on a scale | 1.6 (0.85)

4. Secondary Outcome: Subject Assessment of Appearance and Feel of the Lips Using the Look and Feel Scale
Description: The scale consists of subcategories pertaining to how the subjects perceived aspects of their lips (e.g., softness, smoothness, etc). The outcome measure is the percentage of subjects who scored 0-3 on an 11-point scale, where a lower score on the scale indicates a positive result.
Time Frame: 3 months
Population: All subjects with a Look and Feel assessment
Measure: Number; unit: percentage of subjects
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Number analyzed (Participants) | 60
percentage of subjects
  Lips and Mouth Feel Soft | 72.9
  Lips Feel Smooth | 81.4
  Lips Feel Natural | 93.2
  Lips Look Even | 88.1
  Lips Look Natural | 89.8

5. Secondary Outcome: Number of Subjects Who Attain Their Lip Treatment Goal
Description: Prior to treatment and in consultation with the Investigator, the subject establishes a realistic lip fullness treatment goal. At follow-up, attainment is assessed as yes or no. The outcome measure is the percentage of subjects responding "yes" as to whether their pre-established lip fullness treatment goal had been attained.
Time Frame: 1-12 months
Population: All subjects who provided a lip fullness goal achievement assessment
Measure: Number; unit: percentage of subjects
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Number analyzed (Participants) | 60
percentage of subjects
  Month 1 (n = 58) | 98.3
  Month 3 (n = 59) | 98.3
  Month 6 (n = 59) | 86.4
  Month 9 (n = 59) | 86.4
  Month 12 (n = 58) | 56.9

6. Secondary Outcome: Adverse Events
Time Frame: 12 months
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Number analyzed (Participants) | 60
percentage of subjects
  Bruising | 51.7
  Swelling | 8.3
  Lumps/bumps | 8.3

ADVERSE EVENTS:
Arm/Group | Juvéderm® Ultra Lip Injectable Gel
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 37/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Juvéderm® Ultra Lip Injectable Gel (N=60)
Nerve compression (unrelated to device) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Juvéderm® Ultra Lip Injectable Gel (N=60)
Bruising (General disorders) | 31
Swelling (General disorders) | 5
Lumps/bumps (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.